CLINICAL TRIAL: NCT04896047
Title: Role of FGF19 in Sarcopenia Associated with Chronic Kidney Disease
Brief Title: FGF19 and Chronic Kidney Disease
Acronym: RENAMUS 19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0823
Record Dates: First submitted 2021-03-19; First posted 2021-05-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CKD patients (Experimental): Patients with CKD, non-diabetic, without a history of renal transplantation, without digestive pathology, aged 18 to 70 and an estimate of the glomerular filtration rate (eGFR) <60 ml / min / 1.73m2 according to the formula of CKD-EPI.
  Interventions: Procedure: Meal test and muscle biopsies
- Haemodialysis patients (Active Comparator): Patients on hemodialysis, for more than 3 months, with no history of kidney transplantation, without digestive pathology, aged 18 to 70 with a BMI between 18 and 30 kg / m2
  Interventions: Procedure: Meal test and muscle biopsies
- Healthy volunteers (Active Comparator): Healthy volunteers (controls) recruited from the population of living kidney donors or among patients from the nephrology department whose check-up shows no renal pathology
  Interventions: Procedure: Meal test and muscle biopsies

INTERVENTIONS:
Procedure: Meal test and muscle biopsies — The FGF19 parameters will be assessed in fasting and in postprandial period after the consumption of a hyper-carbohydrate and hyper-lipidic test meal called Flexmeal.
  A muscle biopsies by a needle will be performed before and after the Flexmeal.

SUMMARY:
Sarcopenia in chronic kidney disease (CKD) affects 50% of dialysis patients and 20% of patients with non-dialyzed CKD and reduce quality of life and survival. The pathophysiology of uremic sarcopenia is multifactorial (accumulation of toxins, metabolic disturbances, etc.) and poorly characterized. These pejorative factors are associated with malnutrition and a sedentary lifestyle. Currently, there are no strategies to combat sarcopenia with the exception of physical activity, which is only possible for a limited number of patients due to their comorbidities. Developing new pharmacological strategies to combat sarcopenia is necessary.

FGF19 is a growth factor produced in the ileum involved in metabolic homeostasis. In the laboratory, a new function of FGF19 has been discovered. FGF19 acts as a hormonal factor stimulating muscle mass and strength. Preliminary studies had shown a decrease in the concentration and secretion of FGF19 in response to a meal in haemodialysis patients. However, the link between FGF19, muscle mass and CKD has never been demonstrated. The aim of this study is to assess the relationship between the concentration and secretion of FGF19 and muscle function in a large population of patients with CKD of different stages. Given the hormonal communication between the bone and the muscle, the investigators will also recover the bone histological parameters from a bone biopsy if dialysis patients are to benefit from this as part of their follow-up.

The investigators hypothesize that a decrease in FGF19 concentration and secretion in CKD is associated with a decrease in muscle mass and strength.

ELIGIBILITY:
Inclusion Criteria:

-For the patient population:

* estimated GFR <60 ml / min / 1.73m2 according to the CKD-EPI formula OR patients dialyzed for more than 3 months
* No history of kidney transplant
* BMI between 18 and 30 kg / m²
* For women of childbearing age, at least one method of contraception recognized as effective
* Willing and able to give informed consent

For control group:

* Potential living kidney donor
* Willing and able to give informed consent

For all of the study participants:

o Non diabetic (fasting blood glucose <1.26 g / L, or absence of insulin or oral antidiabetic treatment)

Exclusion Criteria:

* For the patient population:

  * Subjects with a history of colectomy, gut resection or cholecystectomy
  * Having received antibiotics, prebiotics, probiotics in the last 3 months.
  * Taking a high dose laxative treatment (> 2 doses per day) in the last 3 months
  * Hemoglobin <7 g / dl or <9 g / L in case of previous cardiovascular disease
* For control group:

  * DFGe ≤ 80 ml / min / 1.73m2 according to CKD-EPI
  * High blood pressure (PA≥140 / 90 mmHg) or taking antihypertensive treatment
  * Presence of proteinuria (> 0.15 g / 24h) or micro-albuminuria (> 3 mg / mg creatinuria) or hematuria (> 20 GR / mm3)
* For all of the study participants:

  * Hemoglobin <7 g / dl or <9 g / L in case of previous cardiovascular disease
  * Active inflammatory, infectious, cardiovascular or neoplastic disease
  * Period of exclusion from a previous study or already participating in a clinical research protocol having an impact on the study judgment criteria
  * Exposure to ionizing radiation (medical radiological examinations or occupational exposure with exposure greater than 20 mSv) in the 6 months preceding inclusion
  * No affiliation to social security
  * Patient under guardianship or safeguarding justice
  * Pregnant patient (a pregnancy test will be carried out for women of reproductive age o For the patients and control group will accept muscles biopsies
  * Presence of a precarious venous capital that does not allow the placement of a venous catheter - Thrombocytopenia
  * History of arrhythmias or cardiac conduction disorders
  * Taking anticoagulant and / or antiplatelet agent
  * Pulse <50 bpm
  * Allergy to local anesthetics and / or plaster

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2027-02-06 (Estimated); Study Completion 2027-02-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between the fasting plasma concentration of FGF19 and the muscle mass | At the end of the study (55 months)
  Study the correlation between the fasting plasma concentration of FGF19 and the muscle mass in % of body weight, measured by DEXA scanner (Dual-X-Ray-Absorptiometry) in non-dialyzed MRC patients with a measured glomerular filtration rate (mDFG) <60 ml / min /1.73m², hemodialysis patients and healthy voluntary being assessed for a kidney donation or a nephrological check-up with no renal pathology..

SECONDARY OUTCOMES:
Correlation between fasting plasma FGF19 concentration and Glomerular Filtration Rate (GFR) | At the end of the study (55 months)
  Correlation between fasting plasma FGF19 concentration and Glomerular Filtration Rate (GFR) measured by a reference method (Iohexol clearance or Tc DTPA) for non-dialysis patients (in ml/min/1.73m2)
Correlation between fasting plasma FGF19 concentration and muscle strength | At the end of the study (55 months)
  Correlation between fasting plasma FGF19 concentration and muscle strength in kilograms in the Hand Grip
Correlation between fasting plasma FGF19 concentration and muscle performance | At the end of the study (55 months)
  Correlation between fasting plasma FGF19 concentration and muscle performance assessed by the 6-minute walk test (TM6) evaluated in metres and by the SPPB (Short Physical Performance Battery) test with a score between 0 and 12
Correlation between fasting plasma FGF19 concentration and muscle quality | At the end of the study (55 months)
  Correlation between fasting plasma FGF19 concentration and muscle quality assessed by ultrasound (echogenicity intensity (EI) from 0 for black to 255 white and qualitatively by the Heckmatt visual assessment scale (Grade I to IV)).
Correlation between fasting plasma FGF19 concentration and muscle mass | At the end of the study (55 months)
  Correlation between fasting plasma FGF19 concentration and muscle mass obtained by ultrasound by measuring the cross-sectional area (in mm2) of the rectus femoris muscle (RF-CSA, Rectus femoris anatomical cross-sectional area)
Correlation between fasting plasma FGF19 concentration and bone density | At the end of the study (55 months)
  Correlation between fasting plasma FGF19 concentration and bone density determined by DEXA scan (total T-score)
Correlation between fasting plasma FGF19 concentration and bone quality in dialysis patients | At the end of the study (55 months)
  Correlation between fasting plasma FGF19 concentration and bone quality in dialysis patients as assessed by the level of bone remodelling determined on bone biopsy (BFR/BS)
Correlation between fasting plasma FGF19 concentration and physical activity | At the end of the study (55 months)
  Correlation between fasting plasma FGF19 concentration and physical activity assessed by the STAQ questionnaire (in hours/week) only if the primary endpoint is significant.
Correlation between fasting plasma FGF19 concentration and faecal bacterial microbiological profile | At the end of the study (55 months)
  Correlation between fasting plasma FGF19 concentration and faecal bacterial microbiological profile by 16s sequencing of stool samples (analysis performed in a second step)
Correlation between fasting plasma FGF19 concentration and the number of adverse events | At the end of the study (55 months)
  Correlation between fasting plasma FGF19 concentration and the number of adverse events such as mortality, cardiovascular events and fractures throughout the protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon SUD, Pierre-Bénite, France